CLINICAL TRIAL: NCT07327775
Title: Is the Disease Burden of Fibromyalgia Syndrome Higher in Mothers of Children With Attention-Deficit/Hyperactivity Disorder? A Prospective Controlled Study
Brief Title: Fibromyalgia Disease Burden in Mothers of Children With Attention-Deficit/Hyperactivity Disorder
Status: Recruiting | Type: Observational
Sponsor: Sultan 1. Murat State Hospital (Other Government)
Responsible Party: Principal Investigator, Alper Mengi, Associate Professor, Sultan 1. Murat State Hospital
Other Study IDs: 26/11/2025-12/03
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia Syndrome; Disease Burden; Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Fibromyalgia; Attention Deficit Disorder with Hyperactivity | interventions — Cost of Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mothers have children with Attention-Deficit/Hyperactivity Disorder: Mothers with Fibromyalgia Syndrome who have children with Attention-Deficit/Hyperactivity Disorder
  Interventions: Other: Disease Burden
- Mothershave children without psychiatric disorders: Mothers with Fibromyalgia Syndrome who have children without psychiatric disorders
  Interventions: Other: Disease Burden

INTERVENTIONS:
Other: Disease Burden — The demographic characteristics of the participants included in the study-age, educational level, occupation, socioeconomic status, marital status, number of children, and number of children diagnosed with ADHD-will be recorded, and body mass index (BMI) will be calculated.
  The duration of symptoms will be assessed in months. Pain intensity in all patients will be evaluated using the Visual Analog Scale (VAS).
  To assess quality of life and functional status, the Fibromyalgia Impact Questionnaire (FIQ), which has demonstrated validity and reliability in Turkish, will be administered.
  Levels of central sensitization will be assessed using the Central Sensitization Inventory (CSI), which has been validated and shown to be reliable in Turkish.

SUMMARY:
In this study, the investigators aimed to evaluate the impact of having a child diagnosed with Attention-Deficit/Hyperactivity Disorder (ADHD) on parental disease burden in mothers diagnosed with Fibromyalgia Syndrome (FMS).

The study will include 50 mothers with FMS who have a child diagnosed with ADHD and 50 mothers with FMS who have children without any psychiatric disorders.

Among mothers of children followed with a diagnosis of ADHD at the Child and Adolescent Psychiatry Outpatient Clinic of Edirne Sultan 1st Murat State Hospital, the presence of widespread body pain will be assessed. Mothers reporting widespread body pain will be referred to the Pain Management Outpatient Clinic of the same hospital for further evaluation for FMS. Mothers diagnosed with FMS will be included in the study group.

The comparison group will consist of mothers with FMS who have children without any psychiatric disorders. These participants will be selected from patients diagnosed with FMS who present to the Pain Management Outpatient Clinic of Edirne Sultan 1st Murat State Hospital.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Participants with Children Diagnosed with ADHD:

* Being a female aged between 18 and 50 years
* Having one or more children aged 6-17 years diagnosed with Attention Deficit/Hyperactivity Disorder (ADHD) according to DSM-5 diagnostic criteria
* Having a diagnosis of Fibromyalgia Syndrome (FMS according to the 2016 American College of Rheumatology [ACR] criteria)
* Being literate

Inclusion Criteria for Participants with Children Without Psychiatric Disorders:

* Being a female aged between 18 and 50 years
* Having one or more children aged 6-17 years without any psychiatric disorders
* Having a diagnosis of Fibromyalgia Syndrome (FMS) according to the 2016 American College of Rheumatology (ACR) criteria
* Being literate

Exclusion Criteria:

* Receiving regular pharmacological treatment for Fibromyalgia Syndrome
* Having an active psychiatric disorder or using psychiatric medication
* Having a history of infectious disease, chronic inflammatory disease, or malignancy
* Being pregnant or breastfeeding
* Having a central or peripheral nervous system disorder (e.g., cerebrovascular disease, multiple sclerosis)
* Being uncooperative during clinical evaluation
* Having comorbid conditions that may affect quality of life, including congestive heart failure, chronic kidney disease, chronic liver disease, pulmonary disease, uncontrolled diabetes mellitus, or peripheral vascular disease
* Having a diagnosis of hypothyroidism or hyperthyroidism
* Having substance use disorder or alcohol use disorder

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study will include 50 mothers with FMS who have a child diagnosed with ADHD and 50 mothers with FMS who have children without any psychiatric disorders.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
pain severity | Baseline
  Pain intensity in all patients will be assessed using the Visual Analog Scale (VAS). For the VAS assessment, a 10-cm horizontal straight line will be used, where 0 indicates no pain and 10 indicates unbearable pain. The average pain intensity experienced during the previous week will be recorded using the VAS.
quality of life and functional status | Baseline
  To assess quality of life and functional status in patients, the Fibromyalgia Impact Questionnaire (FIQ), which has demonstrated validity and reliability in Turkish, will be used. This questionnaire evaluates 10 domains: physical functioning, overall well-being, work absenteeism, work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety, and depression. The maximum possible score is 100, with higher scores indicating greater functional impairment.
level of central sensitization | Baseline
  Patients' levels of central sensitization will be assessed using the Central Sensitization Inventory (CSI), which has demonstrated validity and reliability in Turkish. The CSI consists of 25 items, each scored on a 5-point Likert scale ranging from 0 to 4. A total score of 40 or higher indicates the presence of central sensitization.

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim Tiryaki, MD, Principal Investigator — Sultan 1. Murat State Hospital
Locations (1):
- Sultan 1. Murat State Hospital, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No